CLINICAL TRIAL: NCT07401797
Title: Specimens for Lung Cancer Panel Design
Status: Recruiting | Type: Observational
Sponsor: Maverix Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: MXDX008
Record Dates: First submitted 2026-02-03; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Lung Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Under 40ml of blood from a single venipuncture or collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Prior cancer: Prior cancer history
- No prior cancer: Indeterminant lung nodules with no prior history of cancer
- Healthy volunteers: Healthy volunteers

SUMMARY:
This is an observational study designed to determine the optimal combination of biomarkers and clinical data for the early detection, confirmation, and better treatment of lung cancer including minimizing recurrence.

DETAILED DESCRIPTION:
Peripheral venous blood and clinical data will be collected from consented subjects with lung nodules identified in radiology that are suspicious for lung cancer before invasive diagnosis or treatment is initiated. Various analyses will be conducted to determine which subset of biomarkers is most likely to be the most useful in the clinic. Attributes considered are accuracy (sensitivity, specificity, improvement over other methods) and ease of collection and transport. Results will not be reported to treating physicians and will not alter care of the patient.

ELIGIBILITY:
6.1 Criteria for the no prior cancer suspicious nodule arm

Inclusion:

1. The patient has at least one indeterminant nodule with a diameter greater than or equal to 5mm and a Mayo SPN risk greater than 5%, identified by radiology, that has not been biopsied or undergone surgery.
2. The patient and the treating physician intend to follow up on the nodule with a biopsy procedure, PET scan, or active surveillance, with the procedure or next surveillance planned within the next 7 months.
3. Ability to understand the study and sign an informed consent form
4. Relevant clinical data accessible
5. Ability and willingness to safely donate 40 mL of blood
6. Ability of the site to collect and process blood per protocol Exclusion

1. The patient has one or more nodules with a Mayo SPN risk over 50% or a diameter of 30mm or greater.

2. The patient has received surgical prep, including antibiotics, anesthesia, etc. Fasting is not exclusionary.

3. Previous cancer diagnosis of any origin. 4. Is currently pregnant 5. Is currently a prisoner or becomes a prisoner at any point during the study 6. Is under age 18, is unable to consent, or requires a different person or entity to consent on their behalf 6.2 Criteria for the previous cancer suspicious nodule arm

Inclusion:

1. The patient has at least one indeterminant nodule with a diameter greater than or equal to 5mm and a Mayo SPN risk greater than 5%, identified by radiology, that has not been biopsied or undergone surgery.

2. The patient and the treating physician intend to follow up on the nodule with a biopsy procedure, PET scan, or active surveillance, with the procedure or next surveillance planned within the next 7 months.

3. The patient has been in remission for a previous cancer not of lung origin for more than 5 years.

4. Ability to understand the study and sign an informed consent form 5. Relevant clinical data accessible 6. Ability and willingness to safely donate 40 mL of blood 7. Ability of the site to collect and process blood per protocol Exclusion

1. The patient has one or more nodules with a Mayo SPN risk over 50% or a diameter of 30mm or greater.
2. The patient has received surgical prep, including antibiotics, anesthesia, etc. Fasting is not exclusionary.
3. Previous cancer diagnosis in the lung (either of lung origin or metastasis to the lung).
4. The treating physician believes the lung nodule is a recurrence of a previously diagnosed cancer.
5. Is currently pregnant
6. Is currently a prisoner or becomes a prisoner at any point during the study
7. Is under age 18, is unable to consent, or requires a different person or entity to consent on their behalf

6.3 Criteria for the healthy volunteer arm

Inclusion:

1. Ability to understand the study and sign an informed consent form
2. Relevant clinical data accessible
3. Ability and willingness to safely donate up to 40 mL of blood
4. The ability of the site to collect and process blood per protocol Exclusion

1. Is currently pregnant 2. Is currently a prisoner or becomes a prisoner at any point during the study 3. Is under age 18, is unable to consent, or requires a different person or entity to consent on their behalf

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals over 18 years old with indeterminate lung nodules identified on CT scans.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-08-07 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Test performance | Two years from final case enrollment
  Analytical validity, clinical validity, and clinical utility. Ability to correctly re-risk indeterminate nodules and ability to change clinical care based on hypothetical treatment plans for different test outcomes. Actual test results will not be provided to physicians, and actual care will not be affected.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Morris, PhD, Principal Investigator — Maverix Medical
Locations (1):
- Maverix Medical, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided
Need to eliminate issues with identifiable information in sequencing data.